CLINICAL TRIAL: NCT07108192
Title: The Effect of Hand Holding and Stress Ball Intervention on Pain and Anxiety During Cataract Surgery: A Randomized Controlled Trial
Brief Title: The Effect of Hand Holding and Stress Ball Intervention on Pain and Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Aysel GUL, Principal Investigator, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-43012747-050.04-489789-435
Record Dates: First submitted 2025-07-24; First posted 2025-08-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cataract Surgery
Keywords: hand holding; stress ball; pain; anxiety; cataract surgery
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stress Ball (Experimental): Non-pharmacological methods are preferred because they are economical, carry minimal risk of complications and can be easily applied in clinical settings. In this context, the stress ball, a distraction method, is effective in providing cognitive focus. Stress ball intevention is reported to be effective on pain, anxiety, satisfaction levels and vital signs of patients.
  Interventions: Other: Stress Ball
- Hand Holding (Experimental): Touch is a critical nursing intervention that conveys empathy. Physical touch is reported to play an important role in calming the patient and showing interest in the patient. It is also reported that physical touch has positive effects on patients' pain, anxiety, satisfaction levels and vital signs. Hand holding is one of the methods of physical touch.
  Interventions: Other: Hand Holding
- Control Group (Active Comparator): Patients do not undergo any additional intervention other than standard routine procedures
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Hand Holding — Hand holding intervention will be performed by the researcher. Before cataract surgery, the researcher will sit in a chair next to the patient and warm his/her hands to a level that does not disturb the patient. 1-2 minutes before cataract surgery, the researcher will hold the patient's hand without gloves, with one hand, with moderate pressure, without rubbing or squeezing it uncomfortably. The hand holding intervention will continue until the cataract surgery is completed
  Arms: Hand Holding
Other: Stress Ball — According to the randomization, the patient in the stress ball group will first be taught the use of stress balls face to face by the researcher. The researcher will place a round, medium-hard, high-quality stress ball of the same brand in the patient's active hand 1-2 minutes before the cataract surgery is started. The patient will be asked to squeeze and relax the stress ball by counting to 5 during cataract surgery. After squeezing the stress ball, he/she should count to 5 and then loosen it. The patient will be asked to continue this process until the cataract surgery is completed.
  Arms: Stress Ball
Other: Control Group — Patients who did not receive any intervention other than standard treatment and care during cataract surgery were defined as the control group.
  Arms: Control Group

SUMMARY:
Cataract surgery is currently primarily performed with topical anesthesia. Although topical anesthesia provides many benefits for patients, they may experience pain, anxiety and discomfort during surgery. It has been reported that increased pain and anxiety during surgery may decrease patient cooperation and satisfaction, making surgery more difficult. In this context, in addition to medical interventions, non-pharmacologic methods are recommended to manage pain and anxiety during surgery. Non-pharmacological methods are reported to be simple, effective and cost-effective. In this context, studies have shown that stress ball application and hand holding are effective strategies for the control of pain and anxiety in patients.

According to this information, the aim of this study was to evaluate the effect of stress ball application and hand holding method used during cataract surgery on patients' pain and anxiety.

Another aim of the study was to determine the effects of stress ball application and hand holding method on patients' satisfaction levels and vital signs.

DETAILED DESCRIPTION:
Cataract is the main cause of visual impairment and blindness globally and surgery remains the only effective treatment for cataract. Today, it is a common procedure for routine cataract surgery under topical anesthesia. Topical anesthesia is most commonly used because it eliminates potential complications such as optic nerve damage, retrobulbar hemorrhage and ocular muscle injury. However, topical anesthesia does not eliminate pain sensitivity of the iris, zonule and ciliary body during cataract surgery. Moreover, patients may experience discomfort due to manipulation of intraocular structures during surgery. However, patients are awake during surgery to follow the surgeon's instructions, which can lead to anxiety and adverse consequences in physiologic parameters such as tachycardia and hypertension. Patients may move during surgery due to anxiety and pain, and may lose visual function due to bleeding or post-surgical complications such as glaucoma. Therefore, assessing and controlling pain and anxiety during surgery is important for patient comfort and surgical prognosis. Moreover, the management of pain and anxiety during surgery not only reduces patients' anxiety but also increases patient cooperation during surgery. In this context, pharmacological as well as non-pharmacological methods are widely used in the management of pain and anxiety. Although the effects of hand holding and stress ball application on patients' pain, anxiety, satisfaction levels and vital signs in various contexts have been reported, their effects, especially during cataract surgery, have not been sufficiently investigated. Therefore, this study aims to contribute to the existing literature by examining the effects of hand holding and stress ball application on patients' pain, anxiety, satisfaction levels and vital signs during cataract and to provide evidence for the importance of the use of nonpharmacologic methods.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* Can understand and speak Turkish
* Clear consciousness, person, place and time oriented
* No hearing and perception problems
* Does not have any mental or neurological disorders that may affect communication (Alzheimer's, dementia, etc.)
* First time cataract surgery
* Those without any psychiatric diagnosis/ treatment (antidepressants, anxiolytics, sedatives, etc.)
* No physical problems in squeezing the stress ball (muscle, joint problems, etc.)
* No analgesic or anesthetic medication 24 hours before the procedure
* Individuals who agree to participate in the study will be included in the study

Exclusion Criteria:

* Conversion of topical anesthesia to general anesthesia during surgery
* A different story of eye surgery
* Hearing, speech, physical or mental disability
* Pregnancy or possible pregnancy
* Those with malignancy
* Taking an analgesic medication at least 24 hours before the procedure
* People with chronic pain
* History of incomplete or canceled cataract procedures
* Hypertension in the patient (>160/100 mmHg)
* Suppurative/infective/inflammatory skin condition of the hands
* Hypersensitivity to touch
* Patients with contact-transmitted diseases
* Being uncomfortable with hand-holding,
* In case of need for emergency intervention by a physician during or immediately after the procedure
* Failure to perform the stress ball application in accordance with the instruction
* Pre-existing neuropathy (muscle joint problem, stroke, etc.)
* Complications during cataract surgery
* Those who want to leave the study voluntarily
* Termination of the procedure due to deterioration of the patient's general condition during the procedure
* Failure to carry out intervention practices in accordance with the determined protocol (Dropping the stress ball during the procedure, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety levels | Anxiety levels of the patients will be evaluated in 2 stages, 15 minutes before surgery and 15 minutes after the surgery is completed.
  Anxiety level of the patients will be evaluated with State Anxiety Inventory Short Version. The short form of the inventory was developed by Zsido and colleagues and adapted to the Turkish population. The form is a 4-point Likert-type inventory consisting of a total of 5 items. Individuals who score 10 and higher on the State Anxiety Inventory Short Version are considered clinically anxious.
Pain levels | Patients' pain levels will be evaluated in 2 stages: intraoperatively and 15 minutes after the operation is completed
  The pain level of the patients will be evaluated by Visual Analog Scale (VAS). Their values range from 0-10. Absence of pain is defined as "0 points" and unbearable pain is defined as "10 points".

SECONDARY OUTCOMES:
Patient satisfaction level | Patients' satisfaction levels will be assessed in a single stage 15 minutes after the operation is completed
  The Visual Analog (VAS) is a valid and reliable tool for measuring subjective feelings such as mood. In this study, it will be used to assess patient satisfaction levels. Their values range from 0-10. High scores on the scale indicate high satisfaction (0=Not at all satisfied, 10=Very satisfied).
Physiological parameters-blood pressure | Patients' blood pressure will be measured 15 minutes before surgery and 15 minutes after surgery is completed.
  systolic and diastolic blood pressure
Physiological parameters-pulse rate | The pulse rate of the patients will be measured 15 minutes before surgery and 15 minutes after surgery is completed.
  Pulse rate
Physiological parameters-respiratory rate | The respiratory rate of the patients will be measured 15 minutes before surgery and 15 minutes after surgery is completed.
  Respiratory rate
Physiological parameters-oxygen saturation | Oxygen saturation of the patients will be measured 15 minutes before surgery and 15 minutes after surgery is completed.
  Oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Aysel GÜL, Phd, Study Director — Sakarya University
Locations (1):
- Yenikent State Hospital, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is planned to be published after the study is completed.